CLINICAL TRIAL: NCT01638663
Title: Effect of Vasopressin Antagonism on Renal Sodium and Water Handling and Circulation During Inhibition of the Nitric Oxide System in Healthy Subjects
Brief Title: Effect of the Aquaretic Tolvaptan on Nitric Oxide System (TORA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, MD, Dr.Sci., Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SAFA-1-2012
Record Dates: First submitted 2012-07-06; First posted 2012-07-12 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Cardiovascular Diseases; Nephropathy
Keywords: Tolvaptan; L-NMMA; Healthy subjects; Nephrology; Cardiology
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan (Active Comparator): Oral administration of 15 mg Tolvaptan on each examination day.
  Interventions: Drug: Tolvaptan
- Placebo (Placebo Comparator): Oral administration of 15 mg Unikalk tablet on each examination day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolvaptan — 15 mg pr day for 1 day
  Other Names: Samsca
  Arms: Tolvaptan
Drug: Placebo — 1 tablet Unikalk 1 pr day for 1 day
  Other Names: Unikalk
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of tolvaptan on renal water, sodium and potassium excretion, plasma concentration of vasoactive hormones,central blood pressure, pulse wave velocity (PWV) and augmentation index, basal and during inhibition of nitric oxide synthesis in healthy subjects.

DETAILED DESCRIPTION:
Tolvaptan is a vasopressin antagonist (V2-antagonist) and is used in treatment of hyponatremia. Animal studies have demonstrated that inhibition of V2 receptors in the renal principal cell increases renal free water clearance and renal sodium excretion.

Treatment with V2-receptor antagonists increases vasopressin concentration in plasma that stimulates V1-receptors in the vascular bed. This may change both central and peripheral hemodynamics and plasma concentration of vasoactive hormones. Changes in hemodynamics and hormone concentration may consequently change renal sodium and water handling.

The nitric oxide system plays a central role in both renal sodium and water handling and regulation of vascular tone and blood pressure.

The effects of tolvaptan the circulation and kidneys is investigated by using measurements of biomarkers specific for the sodium/water balance in the urine and by measurements of vasoactive hormones in the blood after administration of tolvaptan and L-NMMA infusion.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-40 years
* Body Mass Index (BMI) 18,5-30 kg/m2

Exclusion Criteria:

* Anamnestic or clinical signs of heart, lung, lever, kidney and brain disease
* Neoplastic disease
* Drug abuse
* Alcohol abuse
* Medical treatment except peroral anticontraceptive
* Pregnancy
* Smoking
* Abnormal blood and urine sample
* Abnormal ECG
* Blood donation within a month before examination
* Arterial hypertension (>140 mmHg systolic and/or 90 mmHg diastolic)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
CH2O | 5-6 Hours
  Measurement of H2O clearance at baseline, during and after L-NMMA infusion.

SECONDARY OUTCOMES:
Urine biomarkers(Aquaporins, Epithelial Sodium Channels γ and β, Sodium/Chloride and Sodium/Potassium/Chloride cotransporter) | 5-6 Hours
Central blood pressure | 5-6 Hours
Pulse wave velocity | 5-6 Hours
Augmentation Index | 5-6 Hours
Vasoactive Hormones( Angiotensin II, Aldosterone, Endothelin, Atrial Natriuretic Peptide, Brain Natriuretic Peptide, Arginin Vasopressin) | 5-6 Hours
Fractional sodium excretion | 5-6 Hours
  Measurement of Sodium excretion at baseline, during and after L-NMMA infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Safa Therwani, Bachelor, Principal Investigator — Medicinsk Forskning
Locations (1):
- Safa Therwani, Holstebro, Denmark